CLINICAL TRIAL: NCT06289153
Title: Effect of Internal Bracing on Outcomes Following ACL Reconstruction With Quadriceps Tendon: A Randomized Controlled Trial
Brief Title: Internal Bracing Following ACL Reconstruction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not initiated.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-01182
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: ACL Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Internal Brace (Experimental): Patients will undergo ACL Reconstruction (ACLR) with an internal brace. At 6 months post-operation patients will fill out clinical outcome surveys. At the routine 1 year postoperative visit, all patients will fill out clinical outcome surveys and undergo MRI evaluation of the knee.
  Interventions: Device: Arthrex Internal Brace; Procedure: ACL Reconstruction
- Standard ACLR (Active Comparator): Patients will undergo ACLR without an internal brace. At 6 months post-operation patients will fill out clinical outcome surveys. At the routine 1 year postoperative visit, all patients will fill out clinical outcome surveys and undergo MRI evaluation of the knee.
  Interventions: Procedure: ACL Reconstruction

INTERVENTIONS:
Device: Arthrex Internal Brace — The Arthrex Internal Brace method for ACL reconstruction consists of suture tape used to reinforce the ACL during surgery. This suture tape is secured in place with bioabsorbable anchors that gradually degrade within the body over time.
  Arms: Internal Brace
Procedure: ACL Reconstruction — All patients will undergo ACL reconstruction (ACLR) with or without an internal brace.

SUMMARY:
The purpose of this study is to assess Anterior Cruciate Ligament (ACL) healing through analyzing clinical, radiographic, functional and patient-reported outcomes following ACL reconstruction with quadriceps graft with and without internal bracing.

DETAILED DESCRIPTION:
The primary objective is to compare functional outcomes at one year in patients who underwent ACLR with or without internal bracing. The secondary outcomes are to characterize the evidence of ACL healing at 1 year by MRI imaging of the knee and obtain data on clinical and patient reported outcomes at 1 year follow-up.

ELIGIBILITY:
Inclusion Criteria:

• History of ACL injury indicated for isolated reconstruction, without concomitant ligament reconstruction or repair, cartilage repair procedure, or osteotomy.

Exclusion Criteria:

* Patients who underwent concomitant ligament reconstruction or repair, cartilage repair procedure, or osteotomy.
* History of blood-borne diseases including HIV, HBV, HCV, HTLV, and syphilis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-03-26 (Estimated); Study Completion 2026-09-26 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in 2000 International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form at Month 6 Post-Operation | Baseline, Month 6 Post-Operation
  The IKDC is a patient-completed tool assessing knee symptoms (7 items), function (2 items), and sports activities (2 items). Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
Change from Baseline in 2000 IKDC Subjective Knee Evaluation Form Score at Month 12 Post-Operation | Baseline, Month 12 Post-Operation
  The IKDC is a patient-completed tool assessing knee symptoms (7 items), function (2 items), and sports activities (2 items). Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
Change from Baseline in Lysholm Knee Scoring System Score at Month 6 Post-Operation | Baseline, Month 6 Post-Operation
  The Lysholm Knee Scoring System is an 8-item assessment of the prevalence of knee problems. The total score ranges from 0-100; scores between 95 and 100 are regarded as exceptional, 84 and 94 as acceptable, 65 to 83 as fair, and less than 65 as poor.
Change from Baseline in Lysholm Knee Scoring System Score at Month 12 Post-Operation | Baseline, Month 12 Post-Operation
  The Lysholm Knee Scoring System is an 8-item assessment of the prevalence of knee problems. The total score ranges from 0-100; scores between 95 and 100 are regarded as exceptional, 84 and 94 as acceptable, 65 to 83 as fair, and less than 65 as poor.
Change from Baseline in Visual Analogue Scale (VAS) - Pain Score at Month 6 Post-Operation | Baseline, Month 6 Post-Operation
  Participants rate their pain on a scale from 0 (no pain) to 10 (worst pain imaginable); the response is the total score.
Change from Baseline in Visual Analogue Scale (VAS) - Pain Score at Month 12 Post-Operation | Baseline, Month 12 Post-Operation
  Participants rate their pain on a scale from 0 (no pain) to 10 (worst pain imaginable); the response is the total score.

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Gonzalez-Lomas, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
De-identified participant data will not be available to other researchers.